CLINICAL TRIAL: NCT00539916
Title: Effects of Regular and Consequent Citrus Fruit Consumption on Vascular Protection Specific Role of the Component Phytomicronutrients
Brief Title: Effects of Regular and Consequent Citrus Fruits Consumption on Vascular Protection
Acronym: AGRUVASC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Jean Pierre Leroy/Clinical Research and Innovation Director, University Hospital, Bordeaux
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: CHUBX 2007/03
Record Dates: First submitted 2007-10-04; First posted 2007-10-05 (Estimated); Last update posted 2008-08-18 (Estimated); Status verified 2008-08

CONDITIONS: Cardiovascular Disease Risk Factors

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Jus d'orange (Experimental)
  Interventions: Behavioral: Regular orange juice consumption
- Boisson contrôle (Placebo Comparator)
  Interventions: Behavioral: Regular orange juice consumption

INTERVENTIONS:
Behavioral: Regular orange juice consumption — 600 mL /day.

SUMMARY:
Epidemiological studies definitively show that fruit and vegetable consumption is positive for health and more specifically for cardiovascular diseases (CVD) prevention. In France, among fruits, those which are the most frequently consumed are citrus fruits essentially as juices and more specifically as orange juices. However, their health effects have been poorly studied so far. Citrus fruits contain vitamin C associated with various phytomicronutrients i.e. carotenoids (essentially -cryptoxanthin) and polyphenols. Each fruit contains specific compounds: hesperetin in orange, naringenin in grapefruit, eriodyctiol in lemon. Some scientific studies performed either in vitro or in animal models demonstrated properties of these micronutrients which could contribute to a positive health effect of citrus fruits on vascular protection. However data are still missing.

The main goal of this project is to characterize the effect of orange juice consumption on vascular disease risk factors and to evaluate the specific role of their micronutrient compounds (polyphenols and carotenoids) in this protection. To reach this goal, a randomized "cross-over" clinical study will be performed on volunteers presenting a mild hypercholesterolemia. They will consume for 4 weeks an orange juice or a reconstituted drink similar to the orange juice for its composition in carbohydrates, minerals, vitamin C and folates but without phytomicronutrients. The effect of the juice consumption on the vascular function will be monitored exploring lipid abnormalities in plasma, measuring endothelial vasoreactivity (FMD) (Flow Mediated Dilatation), as well as endothelial dysfunction, thrombosis, inflammation and oxidative stress biomarkers in plasma. Comparison of urinary metabolomes after orange juice consumption or that of the reconstituted drink will lead to the identification of the metabolic pathways modulated by the orange juice micronutrients.

Moreover ELISA tests for the two major flavanones from citrus fruits (hesperetin and naringenin) will be developed. They will be used to determine the plasma levels of these molecules in order to analyze the relation "ingested quantity - bioavailable quantity - physiological effect".

The results obtained in this project will allow clarifying citrus fruit effects, and particularly orange juice, in vascular protection.

DETAILED DESCRIPTION:
Scientific context:

Arteriosclerosis is a chronic pathogenic inflammatory-fibro-proliferative process of large and medium-sized arteries that results in the progressive formation of fibrous plaques which in turn, impair the blood flow in vessels. These lesions can either promote an occlusive thrombosis in the affected artery (heart attack, thrombotic stroke) or produce a gradual but relentless stenosis of the arterial lumen. A number of subtle dysfunctions occur at the cellular and molecular levels in the early stages of disease progression associated with the loss of cellular homeostatic functions of endothelial cells, smooth muscle cells and macrophages which constitute the major cell types in the atheroma environment.

Several epidemiological studies shown a negative association between consumption of polyphenol-rich foods (fruits and vegetables) and CVD. This association has been partially explained by the fact that polyphenols interrupt lipid peroxidation which is implicated in the initiation of arteriosclerosis. Polyphenols contribution to the prevention of CVD could be attributable to their antioxidant capacity, hypolipidemic and/or anti-inflammatory properties as well as on their effects on metabolic pathways. Among fruits, citrus fruits are interesting sources of polyphenols (flavanones as glycosides) and carotenoids. A single glass of orange juice may contain between 40 and 140 mg flavanones, which may significantly contribute to the total daily polyphenol intake for the high citrus consumers. The clinical evidence of a role of citrus fruit consumption in the prevention of cardiovascular diseases concerns their hypocholesterolemic effect and the improvement of some biomarkers of oxidative stress, but the specific protective role of the phytomicronutrient provided by these beverages has never been considered. According to the type of citrus, the flavanone molecules are different: hesperetin in orange and clementine, naringenin in grapefruit and eriodyctiol in lemon. These molecules were shown to display antioxidant and hypolipidemic effects. Citrus also contains various carotenoids, like violaxanthin, lutein etc… as well as cryptoxanthin which acts as pro-vitamin A and has a positive role in CVD prevention. The specific health benefits brought by these phytomicronutrients are unknown and a clinical study with specific design to assess the contribution of citrus micronutrients has not been performed yet. Moreover, polyphenols and carotenoids are able to affect the expression of genes involved in atherogenesis. The interaction between these molecules on cellular responses is of particular interest. In fact, they could interplay in the cellular antioxidant network or directly (synergistically or antagonistically) affect gene expression. The unravellings of the mechanisms of regulation of transcriptional control of gene expression seems a promising future line of investigation. Newly developed high throughput technologies make a significant contribution to integrative biology. Studies on phytomicronutrients using the analysis of functional genomics and analysis of phenotypes by metabolic are still in its infancy. Integrated databases are necessary to understand their biological functions. The translation of basic scientific discoveries into applied nutrition is an increasing challenge.

Social and economic context:

CVD in adults are the main cause of morbidity and mortality in Western countries. In France, CVD are responsible for about 170 000 deaths a year i.e. 32% of all deaths, representing a total public heath expenditure estimated to 7.9%. As epidemiological studies show a protective effect of fruit and vegetable consumption towards CVD incidence, the National Programme for Nutrition and Health set up in France advices at least a 400g consumption of fruits and vegetable per day, equivalent to 5 items of crude or cooked fruits or vegetables. The present project will give a solid background for the understanding of the molecular mechanisms of the beneficial effects of polyphenols on human health.

Scientifics and socio-economics goals:

Scientific goals are to clearly establish the effects of phytomicronutrient consumption through orange juice on vascular risk factors. This orange juice intake will take place into a French traditional controlled diet. This means that the project deals with nutritional prevention of one of the major cause of death and health costs in France. It involves one of the most popular sources of citrus fruits. This goal will be reached through an interventional clinical study. The final aim of the present project is to give and diffuse nutritional advices on citrus fruits consumption towards consumers, and to make fruit juices producers aware of the interest to optimize the content of their juices in phytomicronutrients.

Originality and new concepts:

Primary originality of the present project is to focus on the specific contribution of the phyto-micronutrients fraction of citrus (polyphenols and carotenoids) within their natural food matrix to the cardiovascular protection. Such an approach is elicited by conducting a cross over randomized study including in its experimental design a regular intake of orange juice compared to the consumption of a beverage mimicking the composition of orange juice. This control beverage will contain the main nutrients of orange juice (carbohydrates, Vit C, Mg++, K+, folates) except polyphenols and carotenoids. It is now well established that CVD are closely associated with endothelial dysfunction. Thus the present study will focus on the endothelium by evaluating both functional (FMD) and systemic (plasma endothelial biomarkers) parameters.

Selected biochemical parameters are usually measured in clinical studies to demonstrate the metabolic effects of studied nutrients. However, these approaches do not properly deal with the complexity of the interactions occurring between nutrients or with the multiplicity of their biological targets. The metabolic approach offers the novel opportunity to investigate the impact of complex food on the whole physiology of the human organism, through elucidation of subtle but highly significant metabolic changes. The present project will highlight the potentiality of metabolic technology to study the health effects of complex food and dietary patterns in free-living populations.

Disposition of data on micronutrients bioavailability (plasma levels) and biological, biochemical and physiological effects will allow establishing correlation studies between "ingested-circulating-physiological effects".

ELIGIBILITY:
Inclusion Criteria:

* 1.6 < LDL-Cholesterol < 1.9 g/L
* Informed consent signed
* Social security affiliation

Exclusion Criteria:

* Tobacco
* Hypertension
* Diabetes
* Renal or hepatic failure
* Thyroid disease
* Autoimmune disease
* Inflammatory, infectious, or surgical event in the last three months
* Antibiotics, laxative, diuretics
* Vitamins, minerals, polyphenol, carotenoid supplementation in the last three months
* Vegetarian
* Sport : > 5h/week
* High consumption of beverage rich in polyphenols (coffee, wine, fruit juice,...)
* Intestinal disease
* Alcoholism

Ages: 50 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2007-10; Primary Completion 2007-10 (Actual); Study Completion 2008-03 (Actual)

PRIMARY OUTCOMES:
Endothelial function measured by humeral artery vasodilatation technic | At inclusion and at the end of each expirmental period

SECONDARY OUTCOMES:
Lipidic & glycemic balance, Polyphenols & carotenoid plasmatic concentration | At the beginning and the end of each experimental period
Post-prandial lipemia | At the end of each experimental period

CONTACTS AND LOCATIONS:
Overall Officials: Joël CONSTANS, Pr, Principal Investigator — Service de Médecine Interne - Pathologie Vasculaire
Locations (1):
- Hopital Saint André - Service de Médecine Interne - Pathologie Vasculaire, Bordeaux, France

REFERENCES:
- [Background] Hertog MG, Feskens EJ, Hollman PC, Katan MB, Kromhout D. Dietary antioxidant flavonoids and risk of coronary heart disease: the Zutphen Elderly Study. Lancet. 1993 Oct 23;342(8878):1007-11. doi: 10.1016/0140-6736(93)92876-u. PMID 8105262
- [Background] Hertog MG, Kromhout D, Aravanis C, Blackburn H, Buzina R, Fidanza F, Giampaoli S, Jansen A, Menotti A, Nedeljkovic S, et al. Flavonoid intake and long-term risk of coronary heart disease and cancer in the seven countries study. Arch Intern Med. 1995 Feb 27;155(4):381-6. PMID 7848021
- [Background] Knekt P, Jarvinen R, Reunanen A, Maatela J. Flavonoid intake and coronary mortality in Finland: a cohort study. BMJ. 1996 Feb 24;312(7029):478-81. doi: 10.1136/bmj.312.7029.478. PMID 8597679
- [Background] Yochum L, Kushi LH, Meyer K, Folsom AR. Dietary flavonoid intake and risk of cardiovascular disease in postmenopausal women. Am J Epidemiol. 1999 May 15;149(10):943-9. doi: 10.1093/oxfordjournals.aje.a009738. PMID 10342803
- [Background] Geleijnse JM, Launer LJ, Van der Kuip DA, Hofman A, Witteman JC. Inverse association of tea and flavonoid intakes with incident myocardial infarction: the Rotterdam Study. Am J Clin Nutr. 2002 May;75(5):880-6. doi: 10.1093/ajcn/75.5.880. PMID 11976162
- [Background] Leuzzi U, Caristi C, Panzera V, Licandro G. Flavonoids in pigmented orange juice and second-pressure extracts. J Agric Food Chem. 2000 Nov;48(11):5501-6. doi: 10.1021/jf000538o. PMID 11087509
- [Background] Jung HA, Jung MJ, Kim JY, Chung HY, Choi JS. Inhibitory activity of flavonoids from Prunus davidiana and other flavonoids on total ROS and hydroxyl radical generation. Arch Pharm Res. 2003 Oct;26(10):809-15. doi: 10.1007/BF02980025. PMID 14609128
- [Background] Franke AA, Cooney RV, Henning SM, Custer LJ. Bioavailability and antioxidant effects of orange juice components in humans. J Agric Food Chem. 2005 Jun 29;53(13):5170-8. doi: 10.1021/jf050054y. PMID 15969493
- [Background] Lee DH, Gross MD, Jacobs DR Jr; Cardiovascular Risk Development in Young Adults Study. Association of serum carotenoids and tocopherols with gamma-glutamyltransferase: the Cardiovascular Risk Development in Young Adults (CARDIA) Study. Clin Chem. 2004 Mar;50(3):582-8. doi: 10.1373/clinchem.2003.028852. Epub 2004 Jan 15. PMID 14726472
- [Background] Dwyer JH, Paul-Labrador MJ, Fan J, Shircore AM, Merz CN, Dwyer KM. Progression of carotid intima-media thickness and plasma antioxidants: the Los Angeles Atherosclerosis Study. Arterioscler Thromb Vasc Biol. 2004 Feb;24(2):313-9. doi: 10.1161/01.ATV.0000109955.80818.8a. Epub 2003 Dec 1. PMID 14656738
- [Background] Aneja R, Hake PW, Burroughs TJ, Denenberg AG, Wong HR, Zingarelli B. Epigallocatechin, a green tea polyphenol, attenuates myocardial ischemia reperfusion injury in rats. Mol Med. 2004 Jan-Jun;10(1-6):55-62. doi: 10.2119/2004-00032.aneja. PMID 15502883
- [Background] Hadjadj S, Paul JL, Meyer L, Durlach V, Verges B, Ziegler O, Drouin P, Guerci B. Delayed changes in postprandial lipid in young normolipidemic men after a nocturnal vitamin A oral fat load test. J Nutr. 1999 Sep;129(9):1649-55. doi: 10.1093/jn/129.9.1649. PMID 10460199
- [Background] Constans J, Conri C. Circulating markers of endothelial function in cardiovascular disease. Clin Chim Acta. 2006 Jun;368(1-2):33-47. doi: 10.1016/j.cca.2005.12.030. Epub 2006 Mar 10. PMID 16530177
- [Background] Gorinstein S, Caspi A, Libman I, Lerner HT, Huang D, Leontowicz H, Leontowicz M, Tashma Z, Katrich E, Feng S, Trakhtenberg S. Red grapefruit positively influences serum triglyceride level in patients suffering from coronary atherosclerosis: studies in vitro and in humans. J Agric Food Chem. 2006 Mar 8;54(5):1887-92. doi: 10.1021/jf058171g. PMID 16506849
- [Background] Gorinstein S, Leontowicz H, Leontowicz M, Drzewiecki J, Jastrzebski Z, Tapia MS, Katrich E, Trakhtenberg S. Red Star Ruby (Sunrise) and blond qualities of Jaffa grapefruits and their influence on plasma lipid levels and plasma antioxidant activity in rats fed with cholesterol-containing and cholesterol-free diets. Life Sci. 2005 Sep 23;77(19):2384-97. doi: 10.1016/j.lfs.2004.12.049. PMID 15964022
- [Background] Gorinstein S, Leontowicz H, Leontowicz M, Krzeminski R, Gralak M, Delgado-Licon E, Martinez Ayala AL, Katrich E, Trakhtenberg S. Changes in plasma lipid and antioxidant activity in rats as a result of naringin and red grapefruit supplementation. J Agric Food Chem. 2005 Apr 20;53(8):3223-8. doi: 10.1021/jf058014h. PMID 15826081
- [Derived] Constans J, Bennetau-Pelissero C, Martin JF, Rock E, Mazur A, Bedel A, Morand C, Berard AM. Marked antioxidant effect of orange juice intake and its phytomicronutrients in a preliminary randomized cross-over trial on mild hypercholesterolemic men. Clin Nutr. 2015 Dec;34(6):1093-100. doi: 10.1016/j.clnu.2014.12.016. Epub 2014 Dec 26. PMID 25865966